CLINICAL TRIAL: NCT04371523
Title: Hydroxychloroquine to Prevent COVID-19 Disease Amongst Healthcare Workers (PROVIDE): A Parallel Randomized Controlled Trial
Brief Title: Hydroxychloroquine to Prevent COVID-19 Disease Amongst Healthcare Workers
Acronym: PROVIDE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was not initiated due to evidence becoming available that did not support the use of hydroxychloroquine in this population, with potential risk of added harm
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Waleed Al-Hazzani, Intensivist, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3190
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Parallel two-armed, multi-centred, blinded, stratified, superiority, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant, nor the investigators, study coordinators, adjudicator, and data analysts will know if the subject is receiving the hydroxychloroquine or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Hydroxychloroquine (Experimental)
  Interventions: Drug: Apo-Hydroxychloroquine
- Control (Placebo Comparator)
  Interventions: Drug: Matched Placebo

INTERVENTIONS:
Drug: Apo-Hydroxychloroquine — Hydroxychloroquine sulfate 400mg PO BID on day one, then 400mg PO weekly, to be taken with meals for two months total.
  Arms: Intervention - Hydroxychloroquine
Drug: Matched Placebo — Matching Placebo
  Arms: Control

SUMMARY:
The objectives of PROVIDE are to:

1. Determine if prophylactic once weekly hydroxychloroquine reduces the incidence of conversion from SARS-2-CoVnasopharyngeal swab negative to positive
2. To determine if weekly prophylactic hydroxychloroquine reduced the severity of COVID-19 symptoms
3. To determine the safety of taking weekly prophylactic hydroxychloroquine

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older to participate.
* Healthcare workers with primary practice in intensive care unit, general internal medicine,
* COVID-19 testing centres, emergency rooms, and nursing homes.
* COVID_19 symptom free at the time of randomization and have a negative diagnostic swab.

Exclusion Criteria:

* Known COVID-19 positivity defined as: a laboratory confirmed case as defined by the local public health institutes
* Suspected COVID-19 positivity defined as possessing symptoms consistent with COVID-19 infections such as: headache, fever, nausea, vomiting, diarrhea, dyspnea, dry cough
* Healthcare workers with pre-existing retinopathy or serious visual problems
* Healthcare workers with known malignancies receiving active chemotherapy or immune modifying medications
* Healthcare workers with known autoimmune disorders
* Healthcare workers with known QT prolongation
* History of ventricular arrhythmias
* Participants at risk of malignant arrythmias ○ At risk defined as: A sudden loss of consciousness with injury; anyone in their immediate family, under the age of 45year, with sudden cardiac death; anyone family history of long QT syndrome

  * Known sensitivity/allergy to hydroxychloroquine
  * Healthcare workers that are currently pregnant
  * Healthcare workers that are already taking chloroquine or hydroxychloroquine
  * Healthcare workers on colchicine or any other anti-viral medication
  * Healthcare workers taking a medication that may interact with hydroxychloroquine (see table below
  * Inability to take oral medications
  * Inability to provide written consent
  * Known G6PD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Positive for SARS-CoV-2 | 8 weeks
  The number of HCW that tested positive for SARS-CoV-2

SECONDARY OUTCOMES:
Hospital admissions | at any time after first dose to hospital discharge, truncated at 60 days
  The number of HCW that required hospital admission secondary to SARS-CoV-2
Intensive care unit admissions | at any time after first dose to hospital discharge, truncated at 60 days
  The number of HCW that required intensive care unit admission
Intubation and mechanical ventilation | at any time after first dose, truncated at 60 days
  The number of HCW that required intubation and mechanical ventilation
ICU length of stay | from randomization to hospital discharge, truncated at 60 days
  number of days admitted to the ICU
Hospital length of stay | from randomization to hospital discharge, truncated at 60 days
  number of days admitted to the hospital
Mortality | from randomization to 60 days
  Death
Incidence of adverse events | from randomization to 60 days
  Gastrointestinal symptoms (abdominal pain, diarrhea, nausea, vomiting), Hypoglycemia, Abdominal LFTs, Angioedema, Opthalmic (corneal changes, decreased visual acuity, macular degeneration, retinal changes), Bronchospasm

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No